CLINICAL TRIAL: NCT03561545
Title: VISUALIZATION OF THE MICROCIRCULATION IN WEIGHTLESSNESS
Acronym: µGµScan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-096
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional capillary density (Experimental): Functional capillary density during weightlessness
  Interventions: Other: weightlessness (parabolic flight)

INTERVENTIONS:
Other: weightlessness (parabolic flight) — weightlessness (parabolic flight)

SUMMARY:
During weightlessness, the cardiovascular system is subject to rapid changes which has been demonstrated in studies of short term (Space Shuttle) and long term missions to Skylab, MIR, and the International Space Station (Nicogossian et al., 1989; Blomquist, 1994; Platts et al., 2014). There is also evidence for changes in the blood vessel structure, the metabolism and the responses to vasodilator and constrictor substances that might have long-term health consequences resembling the effects of aging on the cardiovascular system (Hughson and Shoemaker, 2004). Cardiovascular adaptations cause an increased incidence of postflight orthostatic intolerance (fainting), decreased cardiac output and reduced exercise capacity. Besides these postflight effects, weightlessness could also have harmful consequences during the flight. For example, it has been shown that cardiac arrhythmia may occur during space missions, even in healthy individuals (Convertino, 2009).

To understand the cardiovascular reactions of the human body to changing conditions of gravity is thus an important aim of space science.

While non-invasive imaging of microcirculation is a very promising tool to evaluate cardiovascular condition, knowledge on the involvement of the microcirculation in cardiovascular alterations induced by weightlessness is very limited and further research in this field seems promising. Before using a non-invasive technique for imaging the microcirculation during space flights, it has to be evaluated on earth.

Different proven simulation models exist for investigating the effects of weightlessness on the human body under terrestrial conditions: head down bed rest, dry and wet immersion, and parabolic flights. Among these models, only parabolic flight recreates a real state of weightlessness (see the participant document of information for a description of parabolic flights). Cardiovascular studies have often been performed during parabolic flights. Within the limitations inherent to the method (short duration of weightlessness - about 21 s - following and followed by hypergravity 20 s periods at 1.8g), some remarkable results have been published over the years.

The aim of our research approach is to test feasibility of the in vivo evaluation of the microcirculation in parabolic flight in order to be able to better describe cardiovascular response mechanisms under these conditions. In this context, we expect alterations in the microcirculatory flow during the weightlessness period of parabolic flight.

Our approach might help develop a diagnostic tool to more easily identify weightlessness-induced cardiovascular diseases and improve strategies for adapting astronauts to weightlessness prior to the space mission.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 67
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women (urine pregnancy test for women of childbearing potential)

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional capillary density | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No